CLINICAL TRIAL: NCT06780007
Title: Effect of Akkermansia Muciniphila Akk11 on Weight Loss in Obese Patients: a Multicenter, Randomized, Double-blind, Placebo-controlled Study.
Brief Title: Weight Loss Effect of Akkermansia Muciniphila in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2025003
Record Dates: First submitted 2025-01-14; First posted 2025-01-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: 28≤BMI≤35Kg/m2
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double(participant, investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): 10B AFU/four capsules/day Akk11, before meals; Storage: store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Four maltodextrin capsules/day, before meals; Storage: store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The trial phase of the study will last 12 weeks and each subject will make 4 follow-up visits (day 0, week 4, week 8 and week 12).
  Arms: Probiotic group
Dietary Supplement: Placebo — The trial phase of the study will last 12 weeks and each subject will make 4 follow-up visits (day 0, week 4, week 8 and week 12).
  Arms: Placebo group

SUMMARY:
This study intends to study the effect of Akkermansia muciniphila on weight loss and the improvement of blood inflammation and metabolic indexes in obese patients with low Body Mass Index (BMI) through multi-center clinical studies, and for the first time to innovatively explore the weight loss mechanism of Akkermansia muciniphila by comparing the changes in brain function and fecal microbiota before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

-

1) Age 18-65 years old; 2）28≤BMI≤35Kg/m2； 3) Willing and able to comply with the protocol during the study period, and be able to cooperate with the completion of various examinations during the trial. Written informed consent is provided prior to entry into study screening, and the patient has understood that the study can be withdrawn at any time from the study without any loss

Exclusion Criteria:

1. Pregnant or lactating women, in the reproductive period and not taking contraceptive measures;
2. Oral antibiotics in the past 1 month prior to enrollment;
3. No use of probiotic prebiotic products before 3 weeks of intervention;
4. people without a fitness fat loss program or history of gastric surgery during the intervention period;
5. Patients with severe gastrointestinal diseases;
6. Those who are known to be allergic to synbiotics or similar products;
7. Patients with no self-awareness and those with mental abnormalities;
8. Have a history of organ transplantation or malignant tumor disease;
9. Concurrent use of other experimental drugs or in other clinical trials;
10. Have a history of alcohol, tobacco and other drug abuse;
11. Those who are expected to be unable to complete the magnetic resonance examination;
12. Combined with serious medical diseases or conditions: such as clinically serious (i.e., active) cardiac disease, severe, uncontrolled medical diseases and infections, severe uncontrollable digestive disorders, severe electrolyte disorders, active disseminated intravascular coagulation, major organ failure, such as decompensated heart, pulmonary, hepatic, renal failure, peripheral neuropathy symptoms, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index(BMI) | Day 0, week4, week8, week12.
  BMI = Weight (kg) / [Height (m)]². 24kg/m² ≤ BMI < 28 kg/m² is in the overweight range, and BMI ≥ 28 kg/m² is in the obesity range.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangpeng Wei, Doctor, Principal Investigator — The First Affiliated Hospital, the Air Force Medical University
Locations (1):
- The First Affiliated Hospital, the Air Force Medical University, Xi'an, Shaanxi, China